CLINICAL TRIAL: NCT04315896
Title: Hydroxychloroquine Treatment for Severe COVID-19 Respiratory Disease: Randomised Clinical Trial (HYDRA Trial)
Brief Title: Hydroxychloroquine Treatment for Severe COVID-19 Pulmonary Infection (HYDRA Trial)
Acronym: HYDRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Respiratory Diseases, Mexico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HidroxycloroquinaCOVID19
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: COVID-19; Severe Acute Respiratory Syndrome
Keywords: COVID-19; Severe acute respiratory syndrome
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Hydroxychloroquine

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Clinical practitioners and data analysts will remain blinded all through the study. Blinding will end in case the attending physician considers the patient should abandon the study or some of the exclusion/elimination criteria apply.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment (Active Comparator): Hydroxychloroquine tablet 200mg every 12 hours for 10 days.
  Interventions: Drug: Hydroxychloroquine
- placebo (Placebo Comparator): identical placebo, one tablet every 12 hours for 10 days
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Hydroxychloroquine — hydroxychloroquine 400mg day for 10 days
  Arms: treatment
Drug: Placebo oral tablet — Placebo oral tablet
  Arms: placebo

SUMMARY:
Double blinded randomized clinical trial designed to evaluate the security and efficacy of hydroxychloroquine as treatment for COVID-19 severe respiratory disease. The investigators hypothesize that a 400mg per day dose of hydroxychloroquine for 10 days will reduce all-cause hospital mortality in patients with severe respiratory COVID-19 disease.

DETAILED DESCRIPTION:
Since hydroxychloroquine is a low cost and safe anti-malaria drug that has proven effects against COVID-19 in vitro. The investigators aim to study the security and efficacy of this drug in trough a double blinded randomized clinical trial. Recruited patients with severe respiratory disease from COVID-19 will be randomized to an intervention group (400mg per day dose of hydroxychloroquine) and placebo. The investigators' main outcome will be all cause hospital mortality. The investigators hypothesize that a 400mg per day dose of hydroxychloroquine for 10 days will reduce all-cause hospital mortality in patients with severe respiratory COVID-19 disease. Results will be compared in an intention to treat analysis. All clinical, analysis and data team members will be blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. negative pregnancy test in women
3. COVID-19 confirmed by rtPCR in any respiratory sample.
4. Severe COVID-19 disease defined as any from the following:

   1. Pulse oximetry less than 91% or a 3% drop from base pulse oximetry or need to increase supplementary oxygen in chronic hypoxia
   2. Need for mechanical ventilation (invasive or non invasive )
   3. Sepsis/septic shock.

Exclusion Criteria:

1. history of anaphylactic shock to hydroxychloroquine.
2. History of previous administration of chloroquine or hydroxychloroquine (within 1 month)
3. decision of attending physician by any reason.
4. History of chronic hepatic disease (Child-Pugh B or C)
5. History of Chronic renal disease (GFR less than 30)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
All-cause hospital mortality | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to120 days
  incidence of all-cause mortality

SECONDARY OUTCOMES:
Length of hospital stay | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to120 days
  Days from ER admission to hospital discharge
Need of mechanical ventilation | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to120 days
  need of invasive or non invasive mechanical ventilation
Ventilator free days | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to120 days
  28 minus days without invasive ventilation support in patients with invasive mechanical ventilation at randomization
Grade 3-4 adverse reaction | From date of randomization until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to120 days
  Adverse Reactions

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Hernandez-Cárdenas, MD. MSc., Principal Investigator — National Institute of Respiratory Diseases - México; Luis-Felipe Jurado-Camacho, MD, Study Director — National Institute of Respiratory Diseases - México; Ireri Thirion-Romero, MD. MSc, Study Chair — National Institute of Respiratory Diseases - México; Sebastian Rodriguez-Llamazares, MD.MPH, Study Chair — National Institute of Respiratory Diseases - México; Rogelio Perez-Padilla, MD. PhD, Study Director — National Institute of Respiratory Diseases - México; Cristobal Guadarrama, MD MSc, Study Chair — National Institute of Respiratory Diseases - México; Joel Vasquez-Pérez, MD, Study Chair — National Institute of Respiratory Diseases - México
Locations (1):
- Instituto Nacional de Enfermedades Respiratorias, "Ismael Cosío Villegas", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
As requested by other investigators.